CLINICAL TRIAL: NCT06193811
Title: Relative Bioavailability of Two Different Tablet Formulations of BI 685509 and Investigation of the Effects of Food and Esomeprazole on the Pharmacokinetics of BI 685509 Following Oral Administration in Healthy Male and Female Subjects (an Open-label, Randomised, Four-way Crossover Trial)
Brief Title: A Study in Healthy People to Compare Two Different Tablets of BI 685509 and to Test How Food and Esomeprazole Influence the Amount of BI 685509 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1366-0042; 2023-506367-33-00 (Other: CTIS)
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: 4-way crossover design within each treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- R-T1-T2-T3 (Experimental): Reference (R): Avenciguat (BI 685509) (TF2), fasted Test 1 (T1): Avenciguat (BI 685509) (iCF), fasted Test 2 (T2): Avenciguat (BI 685509) (iCF), fed Test 3 (T3) Nexium mups from Day -4 to 1; on Day 1 intake of Nexium mups is followed by the intake of Avenciguat (BI 685509) (iCF), fasted There will be a washout period of at least 6 days between Avenciguat (BI 685509) administrations.
  Interventions: Drug: Avenciguat (BI 685509) (intended commercial formulation (iCF)); Drug: Avenciguat (BI 685509) (trial formulation 2 (TF2)); Drug: esomeprazole
- T1-T3-R-T2 (Experimental)
  Interventions: Drug: Avenciguat (BI 685509) (intended commercial formulation (iCF)); Drug: Avenciguat (BI 685509) (trial formulation 2 (TF2)); Drug: esomeprazole
- T2-R-T3-T1 (Experimental)
  Interventions: Drug: Avenciguat (BI 685509) (intended commercial formulation (iCF)); Drug: Avenciguat (BI 685509) (trial formulation 2 (TF2)); Drug: esomeprazole
- T3-T2-T1-R (Experimental)
  Interventions: Drug: Avenciguat (BI 685509) (intended commercial formulation (iCF)); Drug: Avenciguat (BI 685509) (trial formulation 2 (TF2)); Drug: esomeprazole

INTERVENTIONS:
Drug: Avenciguat (BI 685509) (intended commercial formulation (iCF)) — Avenciguat (BI 685509) (intended commercial formulation (iCF))
Drug: Avenciguat (BI 685509) (trial formulation 2 (TF2)) — Avenciguat (BI 685509) (trial formulation 2 (TF2))
Drug: esomeprazole — esomeprazole (Nexium mups)

SUMMARY:
The main objective of this trial is to investigate:

* the relative bioavailability of Avenciguat (BI 685509) TF2 (Reference, R) vs. Avenciguat (BI 685509) iCF (Test 1, T1) tablets under fasted conditions
* the relative bioavailability of Avenciguat (BI 685509) iCF tablets under fasted (T1) and fed (Test 2, T2) conditions
* the relative bioavailability of Avenciguat (BI 685509) iCF tablets given alone (T1) and together with esomeprazole (Test 3, T3) under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12- lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
5. Either male subject, or female subject who meet any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

   * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom
   * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
   * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
   * Sexually abstinent
   * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant
   * Surgically sterilised (including hysterectomy)
   * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to 4 days
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 4 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com